CLINICAL TRIAL: NCT04775030
Title: Methodology for Developing an Occlusal Appliance With CBD Active Carrier
Acronym: CBD-OCC-APP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Aleksandra Nitecka-Buchta, dr n. med., Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBD-OCC-APP
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Temporomandibular Disorder; Myofascial Pain; Cannabis; Electromyography; Occlusal Appliance; CBD
Keywords: Temporomandibular Disorder; Myofascial Pain; Cannabis; Electromyography; Occlusal appliance; CBD
MeSH Terms: conditions — Temporomandibular Joint Disorders; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: experimental and control group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD occlusal appliance (Experimental): CBD occlusal appliance
  Interventions: Drug: CBD occlusal appliance
- occlusal appliance (Placebo Comparator): Traditional material occlusal appliance
  Interventions: Device: Acrylic resin occlusal appliance

INTERVENTIONS:
Drug: CBD occlusal appliance — Occlusal appliance manufactured with CBD molecules released from material to patients oral cavity during sleep time
  Other Names: CBD OCC APP
  Arms: CBD occlusal appliance
Device: Acrylic resin occlusal appliance — Acrylic resin occlusal appliance during sleep time
  Other Names: ACRYLIC OCC APP
  Arms: occlusal appliance

SUMMARY:
Evaluation of the efficacy of the occlusal appliance with active cannabidiol (CBD) molecules in TMD patients

DETAILED DESCRIPTION:
Occlusal appliance therapies are used in TMD patients. In this research the active CBD molecules will be released from the occlusal appliance during nighttime, in population of patients suffering from TMD. The effectiveness of the myorelaxation (sEMG of mastcatory muscles activity) and analgesic effect( VAS analysis) of occlusal appliance with the CBD molecules will be compared to the traditional acrylic-resin material used so far for occlusal appliance manufacture. The aim of the research is the evaluation of the innovative material effectiveness, used for the production of the occlusal appliance.

ELIGIBILITY:
Inclusion Criteria:

* patient agreement to take part in the study
* RDC/TMD group Ia and Ib
* Bruxism Index> 3 ( Brux-off polysomnography)

Exclusion Criteria:

* CBD allergy/hypersensitivity/ addiction
* Therapy with analgesic drugs
* Therapy with drugs affecting muscle function
* Fixed or removable dental prosthesis
* Ongoing orthodontic treatment
* Other general disorders affecting muscle tension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of sEMG activity of masseter muscle | 40 days
  Reduction of sEMG activity of masseter muscle

SECONDARY OUTCOMES:
Reduction of pain intensity in VAS | 40 days
  Reduction of pain intensity in VAS

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Antonowicz, Adiunct, Principal Investigator — Technical University of Silesia
Locations (1):
- Department of TMD Silesian Medical University, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaney C, Heinzel-Gutenbrunner M, Jobin P, Tschopp F, Gattlen B, Hagen U, Schnelle M, Reif M. Efficacy, safety and tolerability of an orally administered cannabis extract in the treatment of spasticity in patients with multiple sclerosis: a randomized, double-blind, placebo-controlled, crossover study. Mult Scler. 2004 Aug;10(4):417-24. doi: 10.1191/1352458504ms1048oa. PMID 15327040
- [Background] Koppel BS, Brust JC, Fife T, Bronstein J, Youssof S, Gronseth G, Gloss D. Systematic review: efficacy and safety of medical marijuana in selected neurologic disorders [RETIRED]: report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2014 Apr 29;82(17):1556-63. doi: 10.1212/WNL.0000000000000363. PMID 24778283
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, Santiago V, Winocur E, De Laat A, De Leeuw R, Koyano K, Lavigne GJ, Svensson P, Manfredini D. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018 Nov;45(11):837-844. doi: 10.1111/joor.12663. Epub 2018 Jun 21. PMID 29926505
- [Background] Nitecka-Buchta A, Nowak-Wachol A, Wachol K, Walczynska-Dragon K, Olczyk P, Batoryna O, Kempa W, Baron S. Myorelaxant Effect of Transdermal Cannabidiol Application in Patients with TMD: A Randomized, Double-Blind Trial. J Clin Med. 2019 Nov 6;8(11):1886. doi: 10.3390/jcm8111886. PMID 31698733